CLINICAL TRIAL: NCT00873990
Title: Split Mouth Clinical Trial of Fissure Sealant Retention With Self Etching and Total Etch Bonding Agent
Brief Title: Fissure Sealant Retention Trial
Acronym: FSRT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Dr Nadia Aman, The Aga Khan University Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 07GS028SUR
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-03

CONDITIONS: Fissure Sealant Loss
Keywords: fissure sealant; self etch; total etch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): application of total etch bonding agent ( 5th generation) for placement of resing based pit and fissure sealants.
  Interventions: Other: Total etch bonding agent (5th generation)
- 2 (Experimental): Self etch bonding agent (7th generation) application for placement of resin based pit and fissure sealant
  Interventions: Other: Self etch (7th generation ) bonding agent

INTERVENTIONS:
Other: Total etch bonding agent (5th generation) — Selected teeth would receive prophylaxis with pumice using prophylaxis brushes for 20 seconds. The teeth will be isolated with cotton rolls before application of bonding agent. The tooth selected for etch and rinse bonding system (two step bonding agent) will be treated with 37% phosphoric acid (Total Etch Ivoclar Vivadent) for 15 seconds followed by rinsing for 30 seconds and then drying with air syringe till frosty white appearance is achieved.
  Adper Single Bond 2 (3M ESPE) will be applied to occlusal fissure using applicator brushes followed by curing for 10 seconds. Clinpro(3M ESPE) fissure sealant will be applied to pits and fissures and then light cured for 20 seconds.
  Other Names: Adper Single bond 3M ESPE
  Arms: 1
Other: Self etch (7th generation ) bonding agent — For teeth selected for application of self etching bonding agent (Adper Easy Bond 3 M), the bonding agent will be applied to occlusal surface with microbrushes and will be left undisturbed for 20 seconds followed by air drying for 5 seconds and then will be light cured for 10 seconds. Fissure sealant (Clinpro 3M ESPE) will be applied in a similar manner as for etch and rinse group and light cured.
  Other Names: Adper Easy bond 3M ESPE
  Arms: 2

SUMMARY:
The aim of the investigators study is to compare how two different bonding agents affects retention in a preventive dental procedure of pit and fissure sealant. This study will help in deciding whether the self etch bonding agent requiring less steps in completion is as effective as the total etch bonding agent requiring multiple steps in fissure sealant placement.

DETAILED DESCRIPTION:
Pit and fissure sealant have been hailed as a highly effective preventive dental treatment since it was introduced first in late 1970s . Sealants have traditionally placed using two step bonding agents based on acid etching with phosphoric acid followed by drying and bonding agent application and curing. Multiple steps in application of bonding agents have been associated with more chances of procedure errors and prolonged procedure time. The newer bonding agents are based on minimizing the number of steps involved with introduction of self etching bonding agents.6th generation adhesives are based on mixing of two components where as the 7th generation adhesives are based on no mix technique.

Previous studies on fissure sealants have focused on conventional etch and rinse bonding agents, there are only few published studies on effectiveness of the self etch bonding agents in retention of fissure sealants in vivo that have targeted the 6th generation adhesive. Feigal and Quelhas reported equivocal results with use of self etching bonding agents in comparison with etch and rinse bonding agents, but their study was limited by smaller sample size. Similar study was conducted by Burbridge which was based on short clinical follow up of 6 month evaluation where Xeno III by Dentsply (6th generation bonding agent) was compared with Prime & Bond (Dentsply). Another study by Venker et al on Adper Prompt L Pop in a school sealant program was based on retrospective review of cases. In light of published literature on (6th generation) self etch bonding agent has been found to be equal or inferior to total etch bonding agents (5th generation). There are no published clinical trials on the retentiong rate comparison of total etch bonding agent with no mix slef etch bonding agents in pit and fissure sealant.

Our study is based on comparison of effectiveness of single step bonding agent (7th generation adhesives) versus two step bonding agent in fissure sealant retention.

ELIGIBILITY:
Inclusion Criteria:

* Fully erupted bilateral first or second permanent molar teeth.
* Patients requiring fissure sealant due high caries risk.
* Age group 6-25 years.
* Occlusal fissures of molar teeth.

Exclusion Criteria:

* Cases where one of the molar on either side is grossly carious or restored
* Third molars
* Uncooperative patients
* Molar teeth with antagonist tooth not present or extracted
* Mentally and physically handicapped patients

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 93 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-07 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
fissure sealant loss | 3months

SECONDARY OUTCOMES:
fissure sealant loss | 6months

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Aman, BDS, Principal Investigator — The Aga Khan University Hospital
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan